CLINICAL TRIAL: NCT01937702
Title: A Trial Investigating the Influence of Injection Speed and Volume on the Perception of Subcutaneous Injection Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: PSIP
Record Dates: First submitted 2013-08-27; First posted 2013-09-09 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-diabetes medication (Experimental): Insulin
  Interventions: Other: 0.9% NaCl (sodium chloride)

INTERVENTIONS:
Other: 0.9% NaCl (sodium chloride)

SUMMARY:
A trial, investigating the influence of injection speed and volume on the perception of subcutaneous injection pain.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the informed consent form prior to screening
* Age 18-74 years at screening (both included)

Exclusion Criteria:

* Known or suspected hypersensitivity to needle, ink ball pen or other that are in contact with the injection area during the clinical visit
* Previous participation in this trial. Participation is defined as having received at least one injection

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
injection pain | within 24 hours after injection

SECONDARY OUTCOMES:
variability of injection pain | within the first 24 hours after injection

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, Prof, MD, Principal Investigator — Profil Mainz GmbH & Co KG
Locations (1):
- Profil Mainz GmbH & Co. KG, Mainz, Rhineland-Palatinate, Germany